CLINICAL TRIAL: NCT01511107
Title: A Phase 2b, Multicenter, Randomized, Double Blind, Placebo-Controlled Clinical Trial to Evaluate the Efficacy of Short-Course Antimicrobial Therapy for Young Children With Acute Otitis Media (AOM) and Impact on Antimicrobial Resistance
Brief Title: Efficacy of Short-Course Antimicrobial Treatment for Children With Acute Otitis Media and Impact on Resistance
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The primary objective of the study was met.
Sponsor: Alejandro Hoberman (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Alejandro Hoberman, Professor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-0083; AI2009058 (Other: NIH NIAID)
Record Dates: First submitted 2012-01-10; First posted 2012-01-18 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Acute Otitis Media
Keywords: acute otitis media; ear infection; antimicrobial therapy; antimicrobial resistance
MeSH Terms: conditions — Otitis Media; Otitis | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxicillin-Clavulanate, 10 days (Active Comparator): amoxicillin-clavulanate, 90/6.4 mg/kg/day, 2 divided doses, 10 days
  Interventions: Drug: Amoxicillin-Clavulanate, 10 days
- Amoxicillin-Clavulanate, 5 days (Other): amoxicillin-clavulanate, 90/6.4 mg/kg/day, 2 divided doses, 5 days plus placebo, 2 divided doses, 5 days
  Interventions: Drug: Amoxicillin-Clavulanate, 5 days

INTERVENTIONS:
Drug: Amoxicillin-Clavulanate, 10 days — Amoxicillin-clavulanate (90/6.4mg/kg/day in 2 divided doses) Days 1-10
  Other Names: augmentin; amox-clav
  Arms: Amoxicillin-Clavulanate, 10 days
Drug: Amoxicillin-Clavulanate, 5 days — Amoxicillin-clavulanate (90/6.4mg/kg/day in 2 divided doses) Days 1-5
  Plus
  Placebo Days 6-10
  Other Names: augmentin; amox-clav
  Arms: Amoxicillin-Clavulanate, 5 days

SUMMARY:
The investigators will study whether, in young children with acute otitis media (AOM), shortening length of antibiotic treatment as a strategy for reducing antimicrobial resistance provides satisfactory clinical outcome. This is a Phase 2b multicenter, randomized, double-blind, placebo-controlled clinical trial in 600 children aged 6 through 23 months comparing the efficacy of consistent reduced-duration antimicrobial treatment (5 days) with that of consistent standard-duration treatment (10 days) for each episode of AOM developing during a single respiratory season (October 1 through May 31).

DETAILED DESCRIPTION:
Eligible subjects will be randomized at the enrollment visit and will have a telephone call in the course of therapy, and a subsequent visit at the end of therapy. Thereafter, they will be followed through the end of the respiratory season, and their parents will be encouraged to bring their child when concerned about a potential recurrence of AOM. At each recurrence subjects will receive the treatment regimen (either standard- or reduced-duration) to which they were randomized at study entry (consistent treatment strategy).

The recruitment of eligible children with AOM of varying degrees of severity from various primary care practices in 2 separate geographic regions, i.e. Western Pennsylvania and Kentucky, representing urban, suburban and rural demographics will enhance generalizability of study findings and encourage translation to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6 through 23 months
2. Have evidence of AOM defined as:

   * recent (within 48 hours) onset of signs and symptoms as described in the Acute Otitis Media - Severity of Symptoms (AOM-SOS) Scale AND a score of ≥3 at the time of enrollment on the AOM-SOS scale
   * middle ear effusion evidenced by the presence of at least 2 of the following:
   * decreased or absent mobility of the tympanic membrane
   * yellow or white discoloration of the tympanic membrane
   * opacification of the tympanic membrane

   AND
   * acute inflammation evidenced by one of the following:
   * 1+ bulging of the tympanic membrane with either intense erythema or otalgia
   * 2+ or 3+ bulging of the tympanic membrane
3. Has received at least 2 doses of pneumococcal conjugate vaccine
4. Parent has provided informed consent

Exclusion Criteria:

1. Toxic appearance [capillary refill >3 seconds, systolic blood pressure <60 mm Hg];
2. Inpatient hospitalization
3. Clinical or anatomical characteristics that might obscure response to treatment (tympanostomy tubes in place, cleft palate, or Down syndrome)
4. Sensorineural hearing loss (unilateral or bilateral)
5. Serious underlying systemic problems that might obscure response to infection (cystic fibrosis, neoplasm, juvenile diabetes)
6. Concomitant infection that would preclude evaluation of the response of the child's AOM to study product (pneumonia, periorbital cellulitis)
7. Acute wheezing exacerbation which may require treatment with systemic corticosteroids
8. Known renal or hepatic dysfunction or insufficiency
9. History of amoxicillin-clavulanate-associated cholestatic jaundice
10. Immune dysfunction or receipt of immunosuppressive therapy; chronic gastrointestinal conditions (i.e., malabsorption, inflammatory bowel disease)
11. Co-medications (systemic corticosteroids, more than one dose of systemic antimicrobial therapy within 96 hours, receipt of any investigational drug or vaccine within 30 days)
12. Hypersensitivity to penicillin, amoxicillin or amoxicillin-clavulanate, or phenylketonuria or known hypersensitivity to aspartame
13. Unable to complete study, or no access to phone
14. Previously enrolled in this study or currently enrolled in another study

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2012-01; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Hoberman, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaikh N, Hoberman A, Paradise JL, Rockette HE, Kurs-Lasky M, Martin JM. Association Between Nasopharyngeal Colonization and Clinical Outcome in Children With Acute Otitis Media. Pediatr Infect Dis J. 2023 Aug 1;42(8):e274-e277. doi: 10.1097/INF.0000000000003956. Epub 2023 Apr 26. PMID 37171965
- [Derived] Hoberman A, Paradise JL, Rockette HE, Kearney DH, Bhatnagar S, Shope TR, Martin JM, Kurs-Lasky M, Copelli SJ, Colborn DK, Block SL, Labella JJ, Lynch TG, Cohen NL, Haralam M, Pope MA, Nagg JP, Green MD, Shaikh N. Shortened Antimicrobial Treatment for Acute Otitis Media in Young Children. N Engl J Med. 2016 Dec 22;375(25):2446-2456. doi: 10.1056/NEJMoa1606043. PMID 28002709
- [Derived] Martin JM, Hoberman A, Paradise JL, Barbadora KA, Shaikh N, Bhatnagar S, Shope T, Block SL, Haralam MA, Kurs-Lasky M, Colborn DK, Green M. Emergence of Streptococcus pneumoniae serogroups 15 and 35 in nasopharyngeal cultures from young children with acute otitis media. Pediatr Infect Dis J. 2014 Nov;33(11):e286-90. doi: 10.1097/INF.0000000000000445. PMID 24911895

RESULTS

PARTICIPANT FLOW:
Groups:
- Amoxicillin-Clavulanate, 10 Days: Amoxicillin-clavulanate administered at a dosage of 90/6.4mg/kg/day in 2 divided doses for 10 days.
- Amoxicillin-Clavulanate, 5 Days: Amoxicillin-clavulanate administered at a dosage of 90/6.4mg/kg/day in 2 divided doses for Days 1-5 followed by placebo in 2 divided doses for Days 6-10.
Period: Overall Study
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Started | 260 (Randomized to the treatment group.) | 260 (Randomized to the treatment group.)
Completed | 238 (Completed - Assessed at a final visit in Sep or at the end of the respiratory season in Apr or May.) | 219 (Completed - Assessed at a final visit in Sep or at the end of the respiratory season in Apr or May.)
Not Completed | 22 | 41
Not completed — Ineligible | 3 | 2
Not completed — Lost to Follow-up | 10 | 19
Not completed — Withdrawal by Subject | 9 | 20

BASELINE CHARACTERISTICS:
Population: 520 children underwent randomization; 260 were randomized to the amoxicillin-clavulante 10 days group and 260 to the amoxicillin-clavulante 5 days, placebo 5 days group. 3 and 2, respectively, were found ineligible after randomization and were withdrawn by the PI. The remaining 257 and 258 participants, respectively, were the basis for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days | Total
Number analyzed (Participants) | 257 | 258 | 515
Age, Customized [Number; unit: participants]
  6-11 months | 129 | 132 | 261
  12-17 months | 80 | 77 | 157
  18-23 months | 48 | 49 | 97
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 123 | 238
  Male | 142 | 135 | 277
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Parents were asked what ethnicity they would use to describe their child.
  Participants
    Hispanic or Latino | 24 | 23 | 47
    Not Hispanic or Latino | 233 | 235 | 468
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Parents were asked what race or races they would use to describe their child.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 7 | 5 | 12
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 110 | 118 | 228
    White | 116 | 110 | 226
    More than one race | 21 | 21 | 42
    Unknown or Not Reported | 3 | 4 | 7
Study Site [Number; unit: participants] — Participating clinical study sites included: Children's Hospital of Pittsburgh (CHP) of University of Pittsburgh Medical Center (UPMC) Primary Care Center - Oakland, CHP of UPMC Emergency Department, Pittsburgh, Pennsylvania (PA); its affiliated University of Pittsburgh Clinical and Translational Science Institute (PittNet) Pediatric Practice-Based Research Network (PBRN) - PittNet North, East, South, City Loop, Pittsburgh, PA and Kittanning, PA; and Kentucky Pediatric/Adult Research (KPAR) and Physicians to Children and Adolescents (PTCA) Bardstown, Kentucky (KY).
  participants
    Children's Hospital of Pittsburgh (CHP) | 163 | 163 | 326
    Children's Community Pediatrics | 47 | 47 | 94
    Kentucky Pediatric and Adult Research | 47 | 48 | 95
Maternal Education [Number; unit: participants] — Parent was asked about the highest level of maternal education. High school graduate or equivalent implies the mother has graduated high school graduate or has a General Education Diploma (GED) or has attended technical school or some college or has an associates degree.
  participants
    Less than high school | 31 | 26 | 57
    High school graduate or equivalent | 150 | 169 | 319
    College graduate | 76 | 62 | 138
    Unknown | 0 | 1 | 1
Type of Health Insurance [Number; unit: participants] — Type of health insurance relates to the child's insurance.
  participants
    Private | 84 | 75 | 159
    Public | 171 | 179 | 350
    None | 2 | 4 | 6
Exposure to Other Children [Number; unit: participants] — Exposed to other children is defined as a being exposed to 3 or more children for 10 or more hours per week or living in a home with at least 3 other children under the age of 18.
  participants
    Not exposed | 109 | 105 | 214
    Exposed | 148 | 153 | 301
Acute Otitis Media Severity of Symptoms (AOM-SOS) Score [Number; unit: participants] — The AOM-SOS scale measures seven discrete items: tugging of ears, crying, irritability, difficulty sleeping, diminished activity, diminished appetite, and fever. Parents are asked to rate these symptoms in comparison with the child's usual state, as "none," "a little," or "a lot," with corresponding scores of 0, 1, and 2. Thus, total scores range from 0 to 14, with higher scores indicating greater severity of symptoms. Children must have at least a total score of 3 at enrollment to qualify for the study.
  participants
    3-5 | 43 | 59 | 102
    6-8 | 75 | 70 | 145
    9-11 | 98 | 95 | 193
    12-14 | 41 | 34 | 75
Mean AOM-SOS Score [Mean (Standard Deviation); unit: AOM-SOS score] — The AOM-SOS scale measures seven discrete items: tugging of ears, crying, irritability, difficulty sleeping, diminished activity, diminished appetite, and fever. Parents are asked to rate these symptoms in comparison with the child's usual state, as "none," "a little," or "a lot," with corresponding scores of 0, 1, and 2. Thus, total scores range from 0 to 14, with higher scores indicating greater severity of symptoms.
  AOM-SOS score | 8.6 (2.9) | 8.2 (3.0) | 8.4 (3.0)
Estimated severity of illness from pain and fever history only [Number; unit: participants] — AOM episodes were categorized as "likely severe" if the parent described the child as having had "a lot" of ear tugging or "a lot" of fever during the preceding 24 hours, else the episode was categorized as "likely nonsevere."
  participants
    Likely nonsevere | 111 | 121 | 232
    Likely severe | 146 | 137 | 283
Laterality of Acute Otitis Media (AOM) [Number; unit: participants]
  Unilateral | 136 | 126 | 262
  Bilateral | 121 | 132 | 253
Degree of Tympanic Membrane Bulging [Number; unit: participants] — If a child has unilateral AOM, the degree of bulging reflects the degree of bulging in the ear with AOM. If a child has bilateral AOM, the degree of bulging reflects the degree of bulging in the ear with the greater level of bulging,
  participants
    Slight | 35 | 45 | 80
    Moderate | 137 | 135 | 272
    Marked | 85 | 78 | 163
Streptococcus Pneumoniae (S pneumoniae) Sensitivity in Nasopharyngeal Cultures [Number; unit: participants] — Susceptibility to penicillin was determined as follows: When minimum inhibitory concentration (MIC) was available , susceptible was defined as MIC <0.1 µg/mL, intermediate as MIC 0.1 to 1 µg/mL, and resistant as MIC >1 µg/mL. When MIC was not available, susceptible was defined as showing oxacillin disk zone size >20 mm, intermediate as zone size 9 to 20 mm, and resistant as zone size ≤8 mm.
  participants
    S pneumoniae absent | 131 | 120 | 251
    S pneumoniae present, susceptible | 84 | 94 | 178
    S pneumoniae present, intermediate | 20 | 28 | 48
    S pneumoniae present, resistant | 21 | 16 | 37
    Unknown, no culture | 1 | 0 | 1
Haemophilus Influenzae (H influenzae) Sensitivity in Nasopharyngeal Cultures [Number; unit: participants] — Susceptible was defined as beta-lactamase-negative and E test MIC ≤1 µg/mL; nonsusceptible was defined as either beta-lactamase-positive or beta-lactamase-negative and E test MIC >1 µg/mL.
  participants
    H influenzae absent | 172 | 197 | 369
    H influenzae present, susceptible | 53 | 37 | 90
    H influenzae present, nonsusceptible | 31 | 24 | 55
    Unknown, no culture | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Distribution of Children Categorized as Treatment Failure (TF) at or Before the Day 12-14 End-of-Treatment Visit Specific to the Index Episode of AOM
Description: Proportion of children initially diagnosed with AOM who experience treatment failure at or before the day 12-14 visit.
  TF is defined as substantial persistence or worsening of symptoms specifically attributable to AOM, or of otoscopic signs of AOM, after 72 hours from the time of randomization, such that additional antimicrobial therapy is deemed advisable. If a parent/legal guardian is unwilling to continue the assigned study product regimen, the participant will be categorized as TF. Should a participant be administered another systemic antibiotic while taking study medication or prior to Day 16, the participant will be considered a TF. Clinical success is defined as complete or substantial resolution of symptoms specifically attributable to AOM for 48 hours and of otoscopic signs of acute inflammation (bulging of the tympanic membrane (TM) or intense erythema), with or without persistence of middle-ear effusion, such that no additional antibiotic therapy is deemed advisable.
Time Frame: From 72 hours after randomization until day 21 of the index episode. The mean day for this visit was 13.2.
Population: The analysis was intent to treat (ITT). The number of participants is equal to the number of children randomized & eligible who had a clinical assessment at or before the day 12-14 visit.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 238 | 229
participants
  Treatment failure | 39 | 77
  Treatment success | 199 | 152
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; The null hypothesis that amoxicillin-clavulanate 5 days, placebo 5 days (reduced duration) is inferior to amoxicillin-clavulanate 10 days (standard duration) is tested against the alternative that reduced duration treatment is noninferior. Assuming failure rates of 15% and 25% in the standard and reduced duration groups, respectively, a 2-sided significance level of .05 and 10% attrition, it was calculated that 300 participants per group, would provide power of 95% for finding inferiority; Test type: Non-Inferiority or Equivalence — A noninferiority margin of 10% was used. Non-inferiority can be established by placing a confidence interval on the difference in the proportion of TFs in subjects randomized to the 10 day regimen and the proportion of TFs in subjects randomized to the 5 day regimen, and determining whether the lower 95% confidence bound is greater than -10%; Difference between proportions = -.172, 95% CI 2-sided [-.253 to -.091], Standard Deviation .039

2. Secondary Outcome: The Distribution of AOM Recurrences Categorized as Treatment Failure (TF) at or Before the Day 12-14 End-of-Treatment Visit
Description: Proportion of AOM recurrences resulting in treatment failure at or before the day 12-14 visit.
  TF is defined as substantial persistence or worsening of symptoms specifically attributable to AOM, or of otoscopic signs of AOM, after 72 hours from the time of the recurrence, such that additional antimicrobial therapy is deemed advisable. If a parent/legal guardian is unwilling to continue the assigned study product regimen, the participant will be categorized as TF. Should a participant be administered another systemic antibiotic while taking study medication or prior to Day 16, the participant will be considered a TF. Clinical success is defined as complete or substantial resolution of symptoms specifically attributable to AOM for 48 hours and of otoscopic signs of acute inflammation (bulging of the TM or intense erythema), with or without persistence of middle-ear effusion, such that no additional antibiotic therapy is deemed advisable.
Time Frame: From 72 hours after the AOM recurrence was diagnosed until day 21 of the recurrence. The mean day for this visit was 13.3.
Population: The analysis was ITT. The number of participants is equal to the number of children randomized & eligible who had a clinical assessment at or before the day 12-14 visit following an AOM recurrence.
Measure: Number; unit: recurrence
Units Other Than Participants: Recurrences
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 101 | 84
Number analyzed (Recurrences) | 133 | 102
recurrence
  Treatment failure | 25 | 29
  Treatment success | 108 | 73
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference between proportions = -.096, 95% CI 2-sided [-.209 to .016], Standard Deviation .053

3. Secondary Outcome: The Distribution of Children With a Nasopharyngeal (NP) Culture at Enrollment That is Negative for AOM Pathogens in Which the Follow-up NP Culture at Day 12-14 Yields a Nonsusceptible Pathogen
Description: AOM pathogens are defined as Streptococcus pneumoniae (S pn) or Haemophilus Influenzae (H flu). In the case of S pn, susceptibility to penicillin was determined as follows: When minimum inhibitory concentration (MIC) was available, susceptible was defined as MIC <0.1 µg/mL, intermediate as MIC 0.1 to 1 µg/mL, and resistant as MIC >1 µg/mL. When MIC was not available, susceptible was defined as showing oxacillin disk zone size >20 mm, intermediate as zone size 9 to 20 mm, and resistant as zone size ≤8 mm. In the case of H flu, susceptible was defined as beta-lactamase-negative and ampicillin E test MIC ≤1 µg/mL; nonsusceptible was defined as either beta-lactamase-positive or beta-lactamase-negative and ampicillin E test MIC >1 µg/mL.
Time Frame: The day 12-14 visit. The mean day for this visit was 13.3.
Population: The analysis was ITT. The participants are randomized & eligible children having a NP culture at enrollment that is negative for both S pn and H flu and a NP culture at the day 12-14 visit which is either positive (+) for >=1 penicillin nonsusceptible pathogen OR pathogen negative (-) or + only for >=1 penicillin susceptible pathogen.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 75 | 72
participants
  + for nonsusceptible pathogen(s) day 12-14 | 15 | 11
  pathogen - or + only for susceptible day 12-14 | 60 | 61
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups in the proportion of children whose NP isolates at enrollment are negative for AOM pathogens for whom the NP culture at day 12-14 yields a nonsusceptible pathogen; Test type: Superiority or Other; p = 0.45, Regression, Logistic

4. Secondary Outcome: The Distribution of AOM Recurrences With a Nasopharyngeal (NP) Culture at Onset That is Negative for AOM Pathogens in Which the Follow-up NP Culture at Day 12-14 Yields a Nonsusceptible Pathogen
Description: as for outcome 3
Time Frame: The day 12-14 visit. The mean day for this visit was 13.4.
Population: The analysis was ITT. The participants are randomized & eligible children having a NP culture at onset that is negative for both S pn and H flu and a NP culture at the day 12-14 visit which is either positive (+) for >=1 penicillin nonsusceptible pathogen OR pathogen negative (-) or + only for >=1 penicillin susceptible pathogen.
Measure: Number; unit: recurrence
Units Other Than Participants: Recurrences
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 42 | 26
Number analyzed (Recurrences) | 46 | 32
recurrence
  + for nonsusceptible pathogen(s) day 12-14 | 12 | 8
  pathogen - or + only for susceptible day 12-14 | 34 | 24
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: For AOM recurrences with a NP culture at onset that is negative for AOM pathogens, there is no difference between the two groups regarding the proportion of NP cultures at Day 12-14 that yield a nonsusceptible pathogen; Test type: Superiority or Other; p = 0.95, Generalized estimating equations

5. Secondary Outcome: The Distribution of Children With a Nasopharyngeal (NP) Culture at Enrollment That is Positive Only for One or More Susceptible Pathogens in Which the Follow-up NP Culture at Day 12-14 Yields a Nonsusceptible Pathogen
Description: as for outcome 3
Time Frame: The day 12-14 visit. The mean day for this visit was 13.2.
Population: The analysis was ITT. The participants are randomized & eligible children having a NP culture at enrollment that is positive only for >=1 susceptible pathogen & a NP culture at the day 12-14 visit which is either positive (+) for >=1 penicillin nonsusceptible pathogen OR pathogen negative (-) or + only for >=1 penicillin susceptible pathogen.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 93 | 90
participants
  + for nonsusceptible pathogen(s) day 12-14 | 10 | 12
  pathogen - or + only for susceptible day 12-14 | 83 | 78
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups in the proportion of children whose NP isolates at enrollment are positive only for one or more susceptible pathogens for whom the NP culture at day 12-14 yields a nonsusceptible pathogen; Test type: Superiority or Other; p = 0.59, Regression, Logistic

6. Secondary Outcome: The Distribution of AOM Recurrences With a Nasopharyngeal (NP) Culture at Onset That is Positive Only for One or More Susceptible Pathogens in Which the Follow-up NP Culture at Day 12-14 Yields a Nonsusceptible Pathogen
Description: as for outcome 3
Time Frame: The day 12-14 visit. The mean day for this visit was 13.9.
Population: The analysis was ITT. The participants are randomized & eligible children having a NP culture at onset that is positive (+) only for one or more susceptible pathogens & a NP culture at the day 12-14 visit which is either + for >=1 penicillin nonsusceptible pathogen OR pathogen negative (-) or + only for >=1 penicillin susceptible pathogen.
Measure: Number; unit: recurrence
Units Other Than Participants: Recurrences
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 39 | 32
Number analyzed (Recurrences) | 44 | 33
recurrence
  + for nonsusceptible pathogen(s) day 12-14 | 8 | 6
  pathogen - or + only for susceptible day 12-14 | 36 | 27
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: For AOM recurrences with a NP culture at onset that is positive only for one or more susceptible pathogens, there is no difference between the two groups regarding the proportion of NP cultures at Day 12-14 that yield a nonsusceptible pathogen; Test type: Superiority or Other; p > 0.99, Generalized estimating equations

7. Secondary Outcome: The Distribution of Children With a Nasopharyngeal (NP) Culture at Enrollment That is Positive for One or More Nonsusceptible Pathogens in Which the Follow-up NP Culture at Day 12-14 Yields a Nonsusceptible Pathogen
Description: as for outcome 3
Time Frame: The end-of-treatment visit. The mean day for this visit was 13.6.
Population: The analysis was ITT. The participants are randomized & eligible children having both a NP culture at enrollment that is positive (+) for one or more nonsusceptible pathogens & a NP culture at the day 12-14 visit which is either + for >=1 penicillin nonsusceptible pathogen OR pathogen negative (-) or + only for >=1 penicillin susceptible pathogen.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 64 | 60
participants
  + for nonsusceptible pathogen(s) day 12-14 | 34 | 28
  pathogen - or + only for susceptible day 12-14 | 30 | 32
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups in the proportion of children whose NP isolates at enrollment are positive for one or more nonsusceptible pathogens for whom the NP culture at day 12-14 yields a nonsusceptible pathogen; Test type: Superiority or Other; p = 0.47, Regression, Logistic

8. Secondary Outcome: The Distribution of AOM Recurrences With a Nasopharyngeal (NP) Culture at Onset That is Positive for One or More Nonsusceptible Pathogens in Which the Follow-up NP Culture at Day 12-14 Yields a Nonsusceptible Pathogen
Description: as for outcome 3
Time Frame: The end-of-treatment visit. The mean day for this visit was 13.4.
Population: The analysis was ITT. The participants are randomized & eligible children having a NP culture at onset that is positive (+) for >=1 nonsusceptible pathogen & a NP culture at the day 12-14 visit which is either + for >=1 penicillin nonsusceptible pathogen OR pathogen negative (-) or + only for >=1 penicillin susceptible pathogen.
Measure: Number; unit: recurrence
Units Other Than Participants: Recurrences
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 29 | 27
Number analyzed (Recurrences) | 33 | 29
recurrence
  + for nonsusceptible pathogen(s) day 12-14 | 17 | 22
  pathogen - or + only for susceptible day 12-14 | 16 | 7
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: For AOM recurrences with a NP culture at onset that is positive for one or more nonsusceptible pathogens, there is no difference between the two groups regarding the proportion of NP cultures at Day 12-14 that yield a nonsusceptible pathogen; Test type: Superiority or Other; p = 0.05, Generalized estimating equations

9. Secondary Outcome: The Distribution of Children Whose Nasopharyngeal (NP) Isolates at Enrollment Are Pathogen Negative or Positive Only for at Least One Susceptible Pathogen Who Become Colonized With Nonsusceptible Pathogens at Any Time Over the Course of Follow-up
Description: as for outcome 3
Time Frame: Day 1 of study entry until day 365
Population: The analysis was ITT. The participants are randomized & eligible children having both a NP culture at enrollment that is either pathogen negative or positive only for >=1 susceptible pathogen and a NP culture at some time over the course of followup.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 181 | 177
participants
  + for a nonsusceptible pathogen during followup | 85 | 78
  - for a nonsusceptible pathogen during followup | 96 | 99
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference in the proportion of subjects whose NP isolates at enrollment are pathogen-negative or positive only for at least one susceptible pathogen who become colonized with penicillin non-susceptible pathogens at any time over the course of follow-up; Test type: Superiority or Other; p = 0.58, Regression, Logistic; The p-value is adjusted for the culture result at enrollment

10. Secondary Outcome: The Distribution of 6 Week Follow-up, Non-Illness Visits During the Respiratory Season at Which a Nonsusceptible Pathogen is Recovered
Description: as for outcome 3
Time Frame: Day 1 of study entry until day 244. The respiratory season is October 1 - May 31, inclusive.
Population: The analysis was ITT. The participants are randomized & eligible children with at least one follow-up, nonillness visit, with a nasopharyngeal (NP) culture which is either positive (+) for >=1 penicillin nonsusceptible pathogens or positive (+) only for >=1 penicillin susceptible pathogens or pathogen negative (-).
Measure: Number; unit: Visit
Units Other Than Participants: Visits
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 211 | 189
Number analyzed (Visits) | 415 | 359
Visit
  + for nonsusceptible pathogen(s) | 79 | 64
  pathogen - or + only for susceptible pathogen(s) | 336 | 295
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference in the proportion of 6 week follow-up, non-illness visits at which a penicillin-nonsusceptible pathogen is recovered; Test type: Superiority or Other; p = 0.74, Generalized estimating equations

11. Secondary Outcome: The Distribution of Children for Whom the Follow-up Nasopharyngeal (NP) Culture at the Day 12-14 Visit, Specific to the Index Episode, Yields a Nonsusceptible Streptococcus Pneumoniae (S pn) Isolate
Description: In the case of S pn, susceptibility to penicillin was determined as follows: When minimum inhibitory concentration (MIC) was available, susceptible was defined as MIC <0.1 µg/mL, intermediate as MIC 0.1 to 1 µg/mL, and resistant as MIC >1 µg/mL. When MIC was not available, susceptible was defined as showing oxacillin disk zone size >20 mm, intermediate as zone size 9 to 20 mm, and resistant as zone size ≤8 mm.
Time Frame: The day 12-14 visit specific to the index episode. The mean day for this visit was 13.4.
Population: The analysis was ITT. The number of participants is equal to the number of children randomized & eligible having a NP culture at the day 12-14 visit following the index episode.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 233 | 222
participants
  S pn, nonsusceptible | 23 | 26
  S pn, susceptible | 5 | 10
  S pn, absent | 205 | 186
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups regarding the proportion of NP cultures at Day 12-14 that yield a nonsusceptible S pn isolate; Test type: Superiority or Other; p = 0.72, Regression, Logistic; The p-value is adjusted for S pn susceptibility at the index episode

12. Secondary Outcome: The Distribution of AOM Recurrences for Which the Follow-up Nasopharyngeal (NP) Culture at the Day 12-14 Visit Yields a Nonsusceptible Streptococcus Pneumoniae (S pn) Isolate
Description: as for outcome 11
Time Frame: The day 12-14 visit following a recurrence. The mean day for this visit was 13.6.
Population: The analysis was ITT. The number of participants is equal to the number of children randomized & eligible having a NP culture at the day 12-14 visit following an AOM recurrence.
Measure: Number; unit: recurrence
Units Other Than Participants: Recurrences
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 100 | 82
Number analyzed (Recurrences) | 131 | 99
recurrence
  S pn, nonsusceptible | 20 | 25
  S pn, susceptible | 4 | 6
  S pn, absent | 107 | 68
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Test type: Superiority or Other; p = 0.05, Generalized estimating equations; The p-value is adjusted for S pn susceptibility at onset of the AOM recurrence

13. Secondary Outcome: The Distribution of Children for Whom the Follow-up Nasopharyngeal (NP) Culture at the Day 12-14 Visit, Specific to the Index Episode, Yields a Nonsusceptible Haemophilus Influenzae (H Flu) Isolate
Description: In the case of H flu, susceptible was defined as beta-lactamase-negative and ampicillin E test MIC ≤1 µg/mL; nonsusceptible was defined as either beta-lactamase-positive or beta-lactamase-negative and ampicillin E test MIC >1 µg/mL.
Time Frame: The day 12-14 visit specific to the index episode. The mean day for this visit was 13.4.
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 233 | 222
participants
  H flu, nonsusceptible | 38 | 28
  H flu, susceptible | 39 | 37
  H flu, absent | 156 | 157
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups regarding the proportion of NP cultures at Day 12-14 that yield a nonsusceptible H flu isolate; Test type: Superiority or Other; p = 0.47, Regression, Logistic; The p-value is adjusted for H flu susceptibility at onset of the index episode

14. Secondary Outcome: The Distribution of AOM Recurrences for Which the Follow-up Nasopharyngeal (NP) Culture at the Day 12-14 Visit Yields a Nonsusceptible Haemophilus Influenzae (H Flu) Isolate
Description: as for outcome 13
Time Frame: The day 12-14 visit following a recurrence. The mean day for this visit was 13.6.
Population: as for outcome 12
Measure: Number; unit: recurrence
Units Other Than Participants: Recurrences
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 100 | 82
Number analyzed (Recurrences) | 131 | 99
recurrence
  H flu, nonsusceptible | 19 | 15
  H flu, susceptible | 17 | 20
  H flu, absent | 95 | 64
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Test type: Superiority or Other; p = 0.69, Generalized estimating equations; The p-value is adjusted for H flu susceptibility at onset of the AOM recurrence

15. Secondary Outcome: The Distribution of Children With AOM Recurrences and Relapses Within 60 Days of Enrollment
Description: An episode of AOM occurring after Day 16 will be considered a recurrence. Subjects seen after day 10 and categorized as clinical success who return for an interim/sick visit before day 17 and are found to have AOM will be categorized as a relapse. For secondary outcome analyses, relapses are combined with recurrences.
Time Frame: Day 1 of study entry until day 60.
Population: The analysis was ITT. The participants are randomized & eligible children having follow-up greater than or equal to day 60.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 241 | 224
participants
  # cumulative recurrences/relapses = 0 | 173 | 173
  # cumulative recurrences/relapses = 1 | 66 | 48
  # cumulative recurrences/relapses = 2 | 2 | 3
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups in the proportion of children followed greater than 60 days having at least one AOM relapse or recurrence within 60 days of enrollment; Test type: Superiority or Other; p = 0.16, Regression, Logistic; The p-value is adjusted for site & the stratification variables, namely age group & exposure or nonexposure to ≥3 children for ≥10 hours per week

16. Secondary Outcome: The Distribution of Children With AOM Recurrences and Relapses Within the Entire Respiratory Season
Description: as for outcome 15
Time Frame: Day 1 of study entry until day 244. The respiratory season is October 1 - May 31, inclusive.
Population: The analysis was ITT. The participants are randomized & eligible children completing the study.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 238 | 219
participants
  # cumulative recurrences/relapses = 0 | 135 | 133
  # cumulative recurrences/relapses = 1 | 61 | 59
  # cumulative recurrences/relapses = 2 | 31 | 20
  # cumulative recurrences/relapses = 3 | 8 | 4
  # cumulative recurrences/relapses = 4 | 3 | 3
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups in the proportion of children completing the study having at least one AOM relapse or recurrence within the entire respiratory season; Test type: Superiority or Other; p = 0.32, Regression, Logistic; [statistical method as in outcome 15, analysis 1]

17. Secondary Outcome: The Mean Rate, Per Month, of Protocol AOM Recurrences and Relapses Within 60 Days of Enrollment
Description: An episode of AOM occurring after Day 16 will be considered a recurrence. Subjects seen after day 10 and categorized as clinical success who return for an interim/sick visit before day 17 and are found to have AOM will be categorized as a relapse. For secondary outcome analyses, relapses are combined with recurrences.
  The rate, expressed as a monthly rate, is calculated by dividing the total number of recurrences and relapses within 60 days of enrollment by the number of months of follow-up within 60 days of enrollment.
Time Frame: Day 1 of study entry until day 60.
Population: The analysis was ITT. The participants are randomized & eligible children having follow-up beyond day 16.
Measure: Mean (Standard Deviation); unit: recurrences/relapses per month
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 245 | 232
recurrences/relapses per month | 0.15 (0.24) | 0.12 (0.23)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups in the rate of recurrences/relapses within 60 days of enrollment; Test type: Superiority or Other; p = 0.23, Regression, Poisson; [statistical method as in outcome 15, analysis 1]

18. Secondary Outcome: The Mean Rate, Per Month, of Protocol AOM Recurrences and Relapses Within the Entire Respiratory Season
Description: An episode of AOM occurring after Day 16 will be considered a recurrence. Subjects seen after day 10 and categorized as clinical success who return for an interim/sick visit before day 17 and are found to have AOM will be categorized as a relapse. For secondary outcome analyses, relapses are combined with recurrences.
  The rate, expressed as a monthly rate, is calculated by dividing the total number of recurrences and relapses by the number of months of follow-up.
Time Frame: Day 1 of study entry until day 244. The respiratory season is October 1 - May 31, inclusive.
Population: The analysis was ITT. The participants are randomized & eligible children having follow-up beyond day 16.
Measure: Mean (Standard Deviation); unit: recurrences/relapses per months followed
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 245 | 232
recurrences/relapses per months followed | 0.14 (0.18) | 0.12 (0.19)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups in the rate of recurrences/relapses within the entire respiratory season; Test type: Superiority or Other; p = 0.22, Regression, Poisson; [statistical method as in outcome 15, analysis 1]

19. Secondary Outcome: The Mean Number of Days Systemic Antibiotics Were Received During the Entire Respiratory Season
Description: Systemic antibiotics include the study product, Amoxicillin-Clavulanate, dispensed for either 10 or 5 days and various concomitant medications, i.e. Amoxicillin, Amox/Clav, Azithromycin, Cefdinir, Cefpodoxime, Ceftriaxone, Erythromycin, Trimethoprim-Sulfamethoxazole, Omnicef, Augmentin, Azithromycin, Cefazolin, Clarythromycin and Ciprofloxacin.
Time Frame: Day 1 of study entry until day 244. The respiratory season is October 1 - May 31, inclusive.
Population: The analysis was ITT. The number of participants is equal to the number of children randomized & eligible.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 257 | 258
days
  Study product | 14.72 (6.77) | 6.79 (3.01)
  Other systemic antibiotic | 6.19 (9.33) | 7.98 (10.94)
  All systemic antibiotics | 20.91 (12.70) | 14.77 (12.10)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups in the mean number of days a systemic antibiotic was received during the respiratory season; Test type: Superiority or Other; p < .001, Regression, Linear; The p-value is adjusted for site & the stratification variables and for length of follow-up

20. Secondary Outcome: The Mean Acute Otitis Media - Severity of Symptom (AOM-SOS) Scores Days 6 to 14
Description: The AOM-SOS scale measures seven discrete items: tugging of ears, crying, irritability, difficulty sleeping, diminished activity, diminished appetite, and fever. The parent rated each of these symptoms in comparison with the child's usual state, as "none," "a little," or "a lot," with corresponding scores of 0, 1, and 2, and recorded the ratings in a diary. Each set of ratings was summed to obtain an AOM-SOS score as a measure of symptom burden. Total scores range from 0 to 14, with higher scores indicating greater severity of symptoms. For instances in which the participant was declared a treatment failure, scores are included up to, but not including the day of the failure. Otherwise, scores day 6 to day 14 are included.
Time Frame: From day 6 of administration of study product until day 14 for all episodes
Population: The analysis was ITT. The number of participants equals the number of children with at least one AOM-SOS score from day 6 of administration of study product to day 14. The scores were based on diaries completed at home by the child's parent.
Measure: Mean (Standard Deviation); unit: AOM-SOS score
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 234 | 230
AOM-SOS score
  Day 6 | 1.72 (2.14) | 1.64 (2.38)
  Day 7 | 1.46 (2.11) | 1.57 (2.53)
  Day 8 | 1.29 (1.99) | 1.56 (2.38)
  Day 9 | 1.29 (2.10) | 1.41 (2.22)
  Day 10 | 1.12 (1.96) | 1.43 (2.36)
  Day 11 | 1.02 (1.84) | 1.40 (2.27)
  Day 12 | 1.07 (1.83) | 1.25 (2.12)
  Day 13 | 1.15 (1.97) | 1.40 (2.47)
  Day 14 | 1.16 (1.93) | 1.37 (2.39)
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups regarding the symptom burden as measured by the respective mean scores over time; Test type: Superiority or Other; p = 0.07, Generalized estimating equations; The p-value is adjusted for site & the stratification variables, episode, day of the diary and AOM-SOS score at the episode

21. Secondary Outcome: The Distribution of Children for Whom Protocol-Defined Diarrhea (PDD) Was Reported and Associated With Study Product
Description: Protocol-defined diarrhea is defined as the occurrence of three or more watery stools in 1 day or two watery stools daily for 2 consecutive days and is limited to events associated with study product.
Time Frame: Day 1 of administration of study product until day 16 for all episodes
Population: The analysis was ITT. The number of participants equals the number of children randomized and eligible.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 257 | 258
participants
  PDD reported | 78 | 75
  PDD not reported | 179 | 183
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups in the proportion of children for whom PDD was reported; Test type: Superiority or Other; p = 0.70, Regression, Logistic; [statistical method as in outcome 15, analysis 1]

22. Secondary Outcome: The Distribution of Children for Whom Diaper Dermatitis Was Reported and Associated With Study Product
Description: Diaper dermatitis is defined as dermatitis in the diaper area calling for prescription of a topical antifungal agent and is limited to events associated with study product.
Time Frame: Day 1 of administration of study product until day 16 for all episodes
Population: The analysis was ITT. The number of participants equals the number of children randomized and eligible.
Measure: Number; unit: participants
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Number analyzed (Participants) | 257 | 258
participants
  Diaper dermatitis reported | 85 | 87
  Diaper dermatitis not reported | 172 | 171
Statistical Analysis 1: Comparison: Amoxicillin-Clavulanate, 10 Days vs Amoxicillin-Clavulanate, 5 Days; Null hypothesis: There is no difference between the two groups in the proportion of children for whom diaper dermatitis was reported; Test type: Superiority or Other; p = 0.86, Regression, Logistic; [statistical method as in outcome 15, analysis 1]

ADVERSE EVENTS:
Time Frame: Parents were interviewed at each scheduled study visit (Day 1, Day 12-14, Day 16-30, 6 week), at the Day 4-6 phone call, at interim illness visits through May 31st, and at the final September visit to determine if their child had any adverse events.
Description: Staff reviewed child's medical records since their last study visit for any adverse events (AEs). A medical condition that was present at the time that the child was screened was considered baseline and not reported as an AE. If the severity of any pre-existing medical condition increased at any time during the study, it was reported as an AE.
Arm/Group | Amoxicillin-Clavulanate, 10 Days | Amoxicillin-Clavulanate, 5 Days
Serious Adverse Events (participants affected / at risk) | 3/257 | 5/258
Other Adverse Events (participants affected / at risk) | 240/257 | 242/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amoxicillin-Clavulanate, 10 Days (N=257) | Amoxicillin-Clavulanate, 5 Days (N=258)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dehydration (General disorders) | 0 (0) | 1 (1)
Fever of unknown origin (General disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Croup (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amoxicillin-Clavulanate, 10 Days (N=257) | Amoxicillin-Clavulanate, 5 Days (N=258)
Non-protocol acute otitis media (AOM) (Ear and labyrinth disorders) | 44 (48) | 48 (60) — Non-protocol AOM refers to AOM diagnosed by a non-protocol provider and not confirmed by a protocol provider.
Gastroenteritis (Gastrointestinal disorders) | 29 (31) | 27 (28)
Protocol defined diarrhea (Gastrointestinal disorders) | 84 (112) | 91 (105) — Protocol defined diarrhea is defined as 3 watery stools in 1 day or 2 watery stools for each of 2 consecutive days.
Vomiting (Gastrointestinal disorders) | 54 (62) | 51 (61)
Fever (General disorders) | 44 (58) | 42 (45)
Viral illness (General disorders) | 30 (32) | 25 (29)
Conjunctivitis (Infections and infestations) | 37 (40) | 36 (37)
Sinusitis (Infections and infestations) | 12 (12) | 8 (9)
Bronchospasm, acute (Respiratory, thoracic and mediastinal disorders) | 48 (65) | 47 (58) — This includes transient episodes of bronchospasm that did not require treatment, as seen in bronchiolitis.
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 197 (469) | 191 (432)
Diaper dermatitis (Skin and subcutaneous tissue disorders) | 166 (300) | 155 (243)
Rash (Skin and subcutaneous tissue disorders) | 27 (30) | 17 (17) — Rash is defined as urticaria or morbilliform or papular rash.
Viral exanthem (Skin and subcutaneous tissue disorders) | 21 (22) | 24 (30)
Tympanostomy tube placement (Surgical and medical procedures) | 19 (19) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No